CLINICAL TRIAL: NCT00976014
Title: Effects of Long-term Therapy With LDL-lowering Plus HDL Raising on Carotid Intima-media Thickness (CIMT) - Carotid Ultrasound Sub-Study of the Familial Atherosclerosis Study-observational Study
Brief Title: Carotid Ultrasound Sub-Study of the Familial Atherosclerosis Study-observational Study
Acronym: FATS
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Xue-Qiao Zhao, Research Professor of Medicine, Cardiology, University of Washington
Other Study IDs: 30519
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intensive Lipid-lowering therapy: Subjects on intensive long-term lipid lowering therapy (lowering LDL-C plus raising of HDL-C).
- Usual Care: Subjects with Atherosclerosis who have been on conventional "standard of care" treatment.

SUMMARY:
This observational study looks at Carotid Stenosis in two groups of subjects using a non-invasive procedure, B-mode ultrasound.

One group of subjects has had long-term intensive lipid altering therapy (lowering LDL-C plus raising HDL-C). The second group of patients has been on conventional "standard of care" treatment for carotid stenosis.

The study will look at the Carotid Intima-media Thickness (CMIT) in both groups.

Hypothesis: CIMT will differ between the two groups, such that the CIMT will be less in the subjects on intensive lipid altering therapy.

ELIGIBILITY:
Inclusion Criteria:

* Intensive Lipid-lowering Therapy Group: Subjects currently enrolled in the Familial Atherosclerosis Treatment Observational Study.
* Usual Care Group: Subjects who were in the FATS OS Study in the past, but have since quit the study and opted for conventional "standard of treatment".

Exclusion Criteria:

* No past or present participation in the FATS OS Study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects known to have Atheroscloerosis.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2006-12-26 (Actual); Primary Completion 2012-05-09 (Actual); Study Completion 2012-05-09 (Actual)

PRIMARY OUTCOMES:
Carotid Intima-media Thickness | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Xue-Qiao Zhao, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Phan BA, Moore AB, Davis J, Pollan LJ, Neradilek B, Brown BG, Zhao XQ. Prolonged combination lipid therapy is associated with reduced carotid intima-media thickness: a case-control study of the 20-year Familial Atherosclerosis Treatment - Observational Study (FATS-OS). J Clin Lipidol. 2014 Sep-Oct;8(5):489-93. doi: 10.1016/j.jacl.2014.07.004. Epub 2014 Jul 12. PMID 25234561